CLINICAL TRIAL: NCT03588507
Title: Clinical and Radiographic Evaluation of Papilla Preservation Flap With or Without Nanocrystalline Hydroxyapatite Bone Graft for Management of Periodontal Intrabony Defects: A Randomized Controlled Clinical Trial
Brief Title: Clinical and Radiographic Evaluation of PPF With or Without NCHA Bone in Treatment of Intrabony Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa ashraf, resident, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ppfrct
Record Dates: First submitted 2018-06-24; First posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Periodontitis; Periodontal Diseases; Periodontal Pocket; Intrabony Periodontal Defect
Keywords: papilla preservation; modified papilla preservation; simplified papilla preservation; nanocrystalline hydroxyapetite; nanobone graft
MeSH Terms: conditions — Periodontitis; Periodontal Diseases; Periodontal Pocket

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: the records of the study participants will be assigned code numbers and the results will be assessed by a third party . coding will not be broken until all assessment and statistics will be completed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Papilla preservation flap techniques (No Intervention): Papilla preservation flap techniques will be conducted to gain access to the intrabony defects. In the narrow interproximal spaces (≤2 mm), incision with the preservation of the buccal papilla according to the simplified papilla preservation technique will be applied. Whereas, in the wide interdental spaces (>2 mm), the modified papilla preservation technique will be applied. Vertical or horizontal mattress sutures and additional interrupted single sutures will be performed to obtain primary closure of the interdental space.
- PPF+NCHA bone graft substitute (Active Comparator): intervention: papilla preservation flap techniques + nanocrystalline hydroxyapatite bone graft substitute Same surgical techniques and procedures will be performed. Before suturing the flap, nanocrystalline hydroxyapatite bone graft substitute(Dentaurum, Germany) will be placed within the defect up to the existing level of the alveolar crest and care will be taken not to overfill the defect. The mucoperiosteal flaps will be repositioned and secured in place using non-resorbable # 6-0-suturing material. Vertical or horizontal mattress sutures and additional interrupted single sutures will be performed to obtain primary closure of the interdental space.
  Interventions: Combination Product: PPF+NCHA bone graft substitute

INTERVENTIONS:
Combination Product: PPF+NCHA bone graft substitute — nanocrystalline hydroxyapatite bone graft is a a newly developed HA containing about 65% water and 35% nanostructured apatite particles. This gave the nanocrystalline hydroxyapatite bone graft many advantages such as providing a close contact with the surrounding tissues, bioresorbability and extremely high number of nano-sized particles and molecules on the surface .
  Arms: PPF+NCHA bone graft substitute

SUMMARY:
This study is meant to assess clinically and radiographically the possible predictable results regarding the use of nanocrystalline hydroxyapatite bone graft substitute together with papilla preservation flap versus papilla preservation flap alone in the treatment of periodontal intrabony defects. Patients will be randomly assigned to either test or control group. The two groups will be equally prepared for both surgical procedures. Then the decision of which group will receive (PPF techniques + Nanocrystalline hydroxyapatite bone graft) and which will receive (PPF techniques only) will be taken.

DETAILED DESCRIPTION:
Treatment of intrabony defects has been indicated mainly to decrease the residual probing depths and so improve tooth prognosis. However, the rationale behind periodontal regeneration was to decrease the pocket depth, improve clinical attachment level and achieve bone fill of severely compromised tooth. However, application of all regenerative strategies needed to be protected by stable soft tissues to avoid exposure and bacterial contamination. That's why modified and simplified papilla preservation flap techniques were developed to maintain the primary closure of interdental sites. The modified papilla preservation technique was developed in order to achieve and maintain primary closure of the flap and to increase the ability to create space for regeneration in the interdental area. The modified papilla preservation technique could be successfully applied in sites in which the interdental space width is at least 2 mm at the most coronal portion of the papilla and in conjunction with a variety of regenerative materials as bone grafts. When interdental sites were narrower, a different papilla preservation procedure had been proposed, the simplified papilla preservation flap In the past years, different Alloplastic synthetic bone graft materials had shown clinical acceptance in the treatment of periodontal osseous defects.Recently, it has been claimed that there were promising results from using nano-sized ceramics as a class of bone graft substitutes due to their improved osseointegration properties. That's why a synthetic nanocrystalline hydroxyapeptite bone grafting material has been introduced for the augmentation of intrabony defects. This gave the nanocrystalline hydroxyapatite bone graft many advantages such as providing a close contact with the surrounding tissues, bioresorbability and extremely high number of nano-sized particles and molecules on the surface.

ELIGIBILITY:
Inclusion Criteria:

* Patient-related criteria:

  * Patient consulting in the outpatient clinic.
  * Able to tolerate surgical periodontal procedures.
  * Patient ready to perform oral hygiene instructions.
  * Compliance with the maintenance program.
  * Provide informed consent.
  * Accepts the 6 months follow-up period.

Teeth related criteria:

* Mature permanent tooth.
* Tooth with two or three-walled intra-bony defect, CAL ≥ 5mm with intra osseous defect ≥ 3mm.

Exclusion Criteria:

* Patient-related criteria:

  * Medically compromised patients.
  * Pregnant or nursing women.
  * Uncooperative patients.
  * Smokers.

Teeth related criteria:

* Teeth with one wall intra-bony defect.
* Teeth with supra-bony defects.
* Teeth with grade II or III mobility.
* Teeth with proximal carious defects or proximal faulty restorations.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level | 6 months
  Measured from the CEJ to the bottom of the gingival sulcus by William's graduated Periodontal probe in mm

SECONDARY OUTCOMES:
Probing Depth | 6 months
  Measured from the gingival margin to the bottom of the gingival sulcus by William's graduated Periodontal probe in mm
Gingival Recession Depth | 6 months
  Measured from the CEJ to the most apical extension of the gingival margin by William's graduated Periodontal probe in mm
Plaque index | 6 months
  Numerical Scoring system Scores 0,1,2,3 by William's graduated Periodontal probe
Gingival index | 6 months
  Numerical Scoring system Scores 0,1,2,3 by William's graduated Periodontal probe
Linear bone fill | 6 months
  Measured from the CEJ to the deepest part of the intrabony defect using the linear measurement tool of the Digora software

CONTACTS AND LOCATIONS:
Overall Officials: Alaa A Rakha, master, Principal Investigator — Cairo University; Noha A Ghallab, professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Heinz B, Kasaj A, Teich M, Jepsen S. Clinical effects of nanocrystalline hydroxyapatite paste in the treatment of intrabony periodontal defects: a randomized controlled clinical study. Clin Oral Investig. 2010 Oct;14(5):525-31. doi: 10.1007/s00784-009-0325-x. Epub 2009 Aug 13. PMID 19680697
- See also: reference link from PubMed — https://www.ncbi.nlm.nih.gov/pubmed/19680697